CLINICAL TRIAL: NCT02796066
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of TSN2898 Topical Gel for the Treatment of Acne Vulgaris
Brief Title: TSN2898-201 Safety and Efficacy of TSN2898 in the Treatment of Acne Vulgaris
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol not approved
Sponsor: Thesan Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSN2898-201
Record Dates: First submitted 2016-05-26; First posted 2016-06-10 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
Keywords: Acne, topical, SCD-1 inhibitor, moderate, severe
MeSH Terms: conditions — Acne Vulgaris; Lymphoma, Follicular | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vehicle (Placebo Comparator): Vehicle gel
  Interventions: Drug: Vehicle
- Low Dose Active (Experimental): Low Dose of TSN2898
  Interventions: Drug: TSN2898
- Mid Dose Active (Experimental): Mid Dose of TSN2898
  Interventions: Drug: TSN2898
- High Dose Active (Experimental): High Dose of TSN2898
  Interventions: Drug: TSN2898

INTERVENTIONS:
Drug: Vehicle — Applied once a day
  Other Names: Topical gel
  Arms: Vehicle
Drug: TSN2898 — Applied once a day
  Other Names: Topical gel
  Arms: Low Dose Active
Drug: TSN2898 — Applied once a day
  Other Names: Topical gel
  Arms: Mid Dose Active
Drug: TSN2898 — Applied once a day
  Other Names: Topical gel
  Arms: High Dose Active

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of TSN 2898 topical gel in the treatment of moderate to severe acne.

DETAILED DESCRIPTION:
TSN2898 is an inhibitor of stearoyl-CoA desaturase-1 (SCD-1), an enzyme present in sebaceous glands and a key regulatory enzyme in lipogenesis. This study will assess the safety and efficacy of TSN2898 topical gel and matched gel vehicle, applied daily on the face for the treatment of moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 16 to 55 years of age
* Must be diagnosed as having moderate or severe acne vulgaris
* ≥ 20 inflammatory lesions on the face
* ≥ 20 non-inflammatory lesions on the face
* ≤ 3 nodule/cyst acne lesions
* Medically healthy
* Females must be of non-childbearing potential

Exclusion Criteria:

* Systemic therapy with retinoids within six (6) months prior to study start
* Topical use of prescription retinoids within four (4) weeks prior to study start
* Oral antibiotics within four (4) weeks prior to study start
* Topical dapsone, sulfacetamide, benzoyl peroxide, α-hydroxy/glycolic acid and retinol/retinaldehyde-containing products, and topical antibiotics, anti-inflammatory medications and corticosteroids on the face within two (2) weeks prior to study start
* Facial procedures, including lasers, peels, and dermabrasion, within two (2) months prior to study start

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 12 weeks

SECONDARY OUTCOMES:
Non-inflammatory lesion counts | 12 weeks
  Absolute change from Baseline
Absolute change from Baseline for inflammatory plus non-inflammatory lesions | 12 weeks
Percent change from Baseline for inflammatory and non-inflammatory lesions | 12 weeks
Investigator's Global Assessment of Acne Severity Score (IGA) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard Welgus, MD, Study Director — Thesan Pharmaceuticals
Locations (6):
- United States (4):
  - Thesan Site 4, San Diego, California
  - Thesan Site 3, Miami, Florida
  - Thesan Site 6, High Point, North Carolina
  - Thesan Site 5, Johnston, Rhode Island
- Thesan Site 2, Santo Domingo, Dominican Republic
- Thesan Site 1, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: No